CLINICAL TRIAL: NCT06920589
Title: Intervention Toward Knowledge of Human Papillomavirus in Homosexual Males
Brief Title: Human Papilloma Virus Awareness Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Univeristario Benemerita Universidad Autonoma de Puebla (Other)
Collaborators: Francisco Javier Báez Hernández (Unknown)
Responsible Party: Principal Investigator, Jorge Alberto Mayo Abarca, Master in nursing, Hospital Univeristario Benemerita Universidad Autonoma de Puebla
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SIEP/ME/112/2021
Record Dates: First submitted 2025-03-13; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Human Papilloma Virus (HPV)
Keywords: intervention; Knowledge; Homosexual me

STUDY DESIGN:
Intervention Model Description: The "Safe and Protected Sex" intervention program for HPV is based on Fisher and Fisher's (1993) IMB model, using social motivation to promote specific preventive actions. It raises cognitive awareness among homosexual men, enhancing their knowledge and understanding of the benefits of protective measures. The program links HPV prevention information to behavior change, incorporating key details on transmission through a horizontal methodology in nursing consultations. The teaching process builds on individuals' perceptions, knowledge, and past experiences. Through reflective learning in nursing consultations, participants make informed decisions, shaping their understanding. HPV knowledge is seen as an evolving process influenced by beliefs, attitudes, concerns, and misconceptions. The intervention fosters a dialogic awareness process, encouraging critical reflection and motivation for prevention, ultimately aiming to create a lasting impact on personal health behavios
Who Masked: Participant
Masking Description: The participants do not know to which group they belong. A single-blind intervention was determined
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Safe and protected sex intervention group (Experimental): This study used the "Safe and Protected Sex" intervention, adapted and validated from an HIV prevention program to focus on HPV. The intervention consists of a single module with two stages aimed at increasing HPV knowledge by enhancing personal (self-determination) and social (controlled behavior) motivation.
  Module 1: "Nursing Consultation on HPV" This structured, planned process follows Corona and Kaltmeier's (2012) horizontal methodology, promoting self-care through social support and trust in nurse-patient dialogue. The goal is to provide counseling on HPV prevention and responsible sexual behavior while acknowledging participants' prior knowledge.
  Stage 1: 4.21-minute educational video, "HPV Fun Facts," uses persuasive narrative to explain HPV transmission, symptoms, complications, and prevention.
  Stage 2: 45-minute "Friendly Educational Guidance" session uses open-ended questions to explore participants' experiences, clarify misconceptions, and reinforce key information
  Interventions: Behavioral: Safe and Protected Sex" intervention targeting HPV
- Placebo control group (Placebo Comparator): For the QA, the baseline measurement (test) was performed once the participant arrived at the sexual health clinic of the School of Nursing with the use of an electronic device that contained the first link of the QuestionPro® platform; subsequently, the participant was given information related to HPV through the usual methodology (diptych) (See Appendix H) that the health system in Mexico carries out. Finally, the second measurement was performed after reading the diptych with the use of the electronic device and the second link of the QuestionPro® platform, prior to the application of the intervention.
  Interventions: Behavioral: Diptych of the Secretary of Health in Mexico

INTERVENTIONS:
Behavioral: Safe and Protected Sex" intervention targeting HPV — This study used the "Safe and Protected Sex" intervention (Báez et al., 2019), adapted and validated from an HIV prevention program to focus on HPV. The intervention consists of a single module with two stages aimed at increasing HPV knowledge by enhancing personal (self-determination) and social (controlled behavior) motivation.
  Module 1: "Nursing Consultation on HPV" This structured, planned process follows Corona and Kaltmeier's (2012) horizontal methodology, promoting self-care through social support and trust in nurse-patient dialogue. The goal is to provide counseling on HPV prevention and responsible sexual behavior while acknowledging participants' prior knowledge.
  Stage 1: A 4.21-minute educational video, "HPV Fun Facts," uses persuasive narrative to explain HPV transmission, symptoms, complications, and prevention.
  Stage 2: A 45-minute "Friendly Educational Guidance" session uses open-ended questions to explore participants' experiences.
  Arms: Safe and protected sex intervention group
Behavioral: Diptych of the Secretary of Health in Mexico — a brochure is provided with general information about the human papilloma virus in men, including the form of contagion, diagnosis, treatment and the use of condoms for prevention.
  Arms: Placebo control group

SUMMARY:
Intervention aimed at increasing knowledge of the human papillomavirus in homosexual men as a means of preventing sexually transmitted diseases and controlling complications associated with the pathology.

DETAILED DESCRIPTION:
Introduction: The World Health Organization reports a 21% prevalence of Human Papillomavirus (HPV) in men, with rates reaching 93% among homosexual men. This group exhibits specific characteristics, such as high rates of sexually transmitted infections (STIs) due to multiple partners and inconsistent condom use, along with limited knowledge about HPV. The intervention "Safe and Protected Sex", using a horizontal methodology, aims to address this health issue.

Objective: To evaluate the effect of the "Safe and Protected Sex" program on HPV knowledge among homosexual men.

Methodology: A quasi-experimental study with a test-retest design and convenience sampling. The sample size was calculated using n'Query Advisor 4.0, resulting in 20 homosexual men per group (n=40).

ELIGIBILITY:
Inclusion Criteria:

* Males who self-identify as homosexual and/or bisexual.
* Engage in sexual relationships with individuals of the same sex.
* Willing to voluntarily participate in the study.
* Have provided informed consent.

Exclusion Criteria:

* Homosexual and/or bisexual males with a profession related to the healthcare field.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Men who identified themselves as homosexual males were considered to be
Enrollment: 40 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
Knowledge of human papillomavirus | 1 month
  This Spanish-language questionnaire is intended to measure knowledge about HPV. It is structured by 38 questions, distributed in four dimensions: 1) causal agent of HPV (1, 2 and 3); 2) risk factors (4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15); 3) signs and symptoms (16, 17, 18, 19 and 20) and 4) prevention, diagnosis and treatment (21, 22, 23, 24, 25, 26, 27, 28, 29, 30, 31, 32, 33, 34, 35, 36, 37 and 38).
  The structure for answering each of the questions is through a Likert-type scale, where three possible options are presented: A= true, B= false and C= don't know. To obtain the cut-off points of the instrument, percentiles (zero to 100) will be used, where Percentile 1 (P125) = no knowledge, Percentile 2 (P250) = insufficient knowledge, Percentile 3 (P375) = fair knowledge and Percentile 4 (P4100) = adequate knowledge

SECONDARY OUTCOMES:
Personal Motivation | 1 month
  To measure personal motivation (self-determination), the Personal Motivation Questionnaire adapted to the Mexican context. It consists of 13 items, which address the preventive behaviors performed by the homosexual male as a result of an emotional-cognitive process, derived from the values and beliefs related to knowledge of HPV, which are manifested during the nursing consultation, through the intervention "Safe and Protected Sex". The response form is Likert type: 1= Strongly agree, 2=Significantly agree, 3= Agree, 4= Neither agree nor disagree, 5= Disagree, 6= Strongly disagree, 7= Strongly disagree, also the score ranges from 13 to 91 points, however for a better interpretation of the data the values are converted into a scale from 0 to 100, where high scores indicate a higher personal motivation during the nursing consultation.
  The validity of the instrument was through eight experts, which yielded a content validity index
social motivation | 1 month
  To measure social motivation (controlled behavior), the Social Motivation Questionnaire adapted to the Mexican context . It consists of 15 items, which deal with the actions that the homosexual male has derived from the social support perceived during the nursing consultancy with horizontal methodology, granted through the intervention "Safe and Protected Sex" directed towards HPV. The response form is Likert type: 1= Strongly agree, 2= Strongly agree, 3= Agree, 4= Neither agree nor disagree, 5= Disagree, 6= Strongly disagree, 7= Strongly disagree, also the score ranges from 15 to 105 points, however for a better interpretation of the data the values are converted into a scale from 0 to 100, where high scores indicate a higher extrinsic motivation during the nursing consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Baez Hernández, Doctor of nursing science, Study Director — Benemerita Universidad Autonoma de Puebla
Locations (1):
- School of Nursing Benemérita Universidad Autonoma de Puebla, Puebla City, Puebla, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
The study continues in a phase of improvement and replication in different contexts to improve its generalization.

REFERENCES:
- [Background] Jeno LM, Raaheim A, Kristensen SM, Kristensen KD, Hole TN, Haugland MJ, Maeland S. The Relative Effect of Team-Based Learning on Motivation and Learning: A Self-Determination Theory Perspective. CBE Life Sci Educ. 2017 Winter;16(4):ar59. doi: 10.1187/cbe.17-03-0055. PMID 29146665
- [Background] Grov C, Rendina HJ, Breslow AS, Ventuneac A, Adelson S, Parsons JT. Characteristics of men who have sex with men (MSM) who attend sex parties: results from a national online sample in the USA. Sex Transm Infect. 2014 Feb;90(1):26-32. doi: 10.1136/sextrans-2013-051094. Epub 2013 Sep 19. PMID 24052337
- [Background] Cranston RD, Carballo-Dieguez A, Gundacker H, Richardson BA, Giguere R, Dolezal C, Siegel A, KunjaraNaAyudhya RP, Gomez K, Piper JM, Lama JR, McGowan I; MTN-017 Protocol Team. Prevalence and determinants of anal human papillomavirus infection in men who have sex with men and transgender women. Int J STD AIDS. 2019 Feb;30(2):154-162. doi: 10.1177/0956462418797864. Epub 2018 Oct 18. PMID 30336747
- [Background] Barrios MC, Rodriguez LS, Pachon CM, Lugo EA. Educational Intervention on Human Papillomavirus in University Students. Indian J Community Med. 2019 Jul-Sep;44(3):213-216. doi: 10.4103/ijcm.IJCM_247_18. PMID 31602105